CLINICAL TRIAL: NCT04119960
Title: Clinical Validation of InferRead Lung CT.AI
Status: Completed | Type: Observational
Sponsor: Infervision (Industry)
Responsible Party: Sponsor
Other Study IDs: InferRead01
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Aided read with InferRead Lung CT.AI — Radiologists read chest CT scans with the aid of InferRead Lung CT.AI

SUMMARY:
Lung cancer is the second most common cause of cancer-related death in men and women. Early pulmonary nodule screening is an effective means to prevent lung cancer, which is no less important than the diagnosis and treatment of lung cancer. Early lung cancer screening has been investigated and applied as a medical practice. InferRead Lung CT.AI by Infervision is a dedicated post processing application that generates CADe marks as an overlay on the original CT series intended to aid the radiologist in the detection of pulmonary nodules. This study was designed to evaluate radiologists' performance in detecting actionable nodules on chest CT when aided by InferRead.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer screening eligible patients

Exclusion Criteria:

-

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung cancer screening eligible patients
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Detection accuracy | 20 hours
  The primary objective of this clinical study is to demonstrate that a radiologist review of a CT scan aided with InferRead Lung CT.AI significantly improves detection of actionable lung nodules. Area under the ROC curve, Sensitivity, specificity, PPV, NPV will be reported, compared between unaided and aided reads.

SECONDARY OUTCOMES:
Reading time change | 20 hours
  The secondary objective of this clinical study is to demonstrate that the radiologist's review time is not significantly increased when aided with InferRead Lung CT.AI. The reading time for each case will be recorded in both aided and unaided reads. The reading times will be compared using a paired T test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States